CLINICAL TRIAL: NCT03112421
Title: Method and Sample Comparison Study of Minicare BNP at a Central Laboratory
Brief Title: Method and Sample Comparison Study Minicare BNP - COMP-BNP-CE03-AN2016
Status: Completed | Type: Observational
Sponsor: Philips Handheld Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: HHDx-07952
Record Dates: First submitted 2017-04-03; First posted 2017-04-13 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure
Keywords: IVD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sample Comparison The objective of this study is to compare the Philips Minicare BNP test with the Centaur BNP test. BNP level measured in human blood samples (EDTA venous whole blood and/or EDTA plasma) will be assessed. Matrix Comparison To compare BNP measurements obtained using Minicare System for EDTA whole blood and EDTA plasma samples.Prior to the study start, a proficiency study will be performed on the Minicare BNP, Architect and I-STAT BNP assay to be sure that devices are performing according to expectations. Approximately 100 EDTA patient whole blood samples covering the entire measuring range of Minicare BNP from LOQ until end of measuring range (expected to be approximately 5000 ng/L) (Ref 7) will be tested (according to CLSI EP09A3 (Ref 5)) at a central laboratory using the Minicare BNP, Alere BNP, I-STAT BNP system. The outcome of the site routine assay (Centaur BNP systems) will be used to evaluate if the blood samples cover the entire distribution range of the assay. If necessary, up to 20% of the samples may be spiked so that the entire range of the assay is covered. The central laboratory will identify the blood tubes with a BNP request. Approximately 1000 μl EDTA whole blood will be available (left over material) for testing on the non-routine devices (i.e., Minicare BNP, Alere BNP, and I-STAT BNP). Testing for the Alere BNP, I-STAT BNP, and Centaur BNP systems will be performed according to the respective IFU's (Ref 1, 2, 3, 4). For the Minicare BNP system, test will be performed according to a DRAFT IFU or a similar document describing the sample treatment and handling for the Minicare BNP system. Alere BNP, I-STAT BNP and Minicare BNP samples should be tested within 6 hours after collection and Centaur BNP samples within 8h of collection. Although different stability claims for BNP, it is highly recommended to perform all measurements on all systems within 2 hours. For Alere BNP, I-STAT BNP, Centaur BNP analysis will be performed using a single blood sample for each patient. Alere BNP and I-STAT will use EDTA whole blood samples as sample type Centaur BNP will be tested on EDTA plasma samples. For the Minicare BNP, both EDTA whole blood and EDTA plasma will be tested for each patient. For the Minicare BNP system the whole blood samples will be tested using a pipette and the same sample will be tested using the SmearSafe Blood Dispenser (transfer device) to investigate a reliable use of such transfer device.

Only the routine Centaur BNP outcomes will be used as part of support for patient diagnosis.

ELIGIBILITY:
Left over blood samples from eligible patients with BNP requests, available at the test site CENTRAL LABORATORY will be selected for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Left over blood samples from eligible patients with BNP requests, available at the test site Central laboratory
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
To investigate the bias between the Philips Minicare BNP test with the Centaur BNP test of the measurement procedures.BNP level measured in human blood samples (EDTA venous whole blood and/or EDTA plasma) will be assessed. | May 2017
  To investigate the bias between the Philips Minicare BNP test with the Centaur BNP test using values spanning the common measuring interval of the measurement procedures.BNP level measured in human blood samples (EDTA venous whole blood and/or EDTA plasma) will be assessed.
To compare BNP measurements obtained using Minicare System for EDTA whole blood and EDTA plasma samples. | May 2017
  To compare BNP measurements obtained using Minicare System for EDTA whole blood and EDTA plasma samples.

SECONDARY OUTCOMES:
Percentage of agreement systems | May 2017
  To estimate the percent of agreement between the Minicare System and three commercially available BNP systems (i.e., Alere BNP, I-STAT BNP, and Centaur BNP tests) using a cut-off value of 100ng/L.
Percentage of agreement samples | May 2017
  To estimate the percent of agreement between EDTA whole blood and EDTA plasma samples for Minicare system using a BNP cut off value of 100ng/L
Evaluate performance of the SmearSafe Blood Dispenser (transfer device), for transferring whole blood from the blood tube directly to the Minicare BNP cartridge. | May 2017
  Evaluate performance of the SmearSafe Blood Dispenser (transfer device), for transferring whole blood from the blood tube directly to the Minicare BNP cartridge, so without use of pipette.

CONTACTS AND LOCATIONS:
Locations (1):
- Diagnostiek voor U, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data that come out of study may be used to publish.